CLINICAL TRIAL: NCT06027606
Title: Cardiovascular Consequences of Prolonged Inhaled Short-acting Beta-agonist Use in Healthy Participants
Brief Title: Cardiovascular Consequences of Inhaled Short-acting Beta-agonist Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00126438
Record Dates: First submitted 2023-08-09; First posted 2023-09-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Albuterol; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Salbutamol (Experimental): Participants are healthy and between the ages of 18-40 years old
  Interventions: Drug: Salbutamol 400mcg
- Budesonide-formoterol (Experimental): Participants are healthy and between the ages of 18-40 years old
  Interventions: Drug: Budesonide/formoterol
- Placebo (Sham Comparator): Participants are healthy and between the ages of 18-40 years old
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol 400mcg — Salbutamol is a short-acting beta-agonist used primarily as a rescue inhaler for respiratory disease such as asthma
  Arms: Salbutamol
Drug: Budesonide/formoterol — Budesonide/formoterol is a inhaled corticosteroid with long-acting beta-agonist component primarily used as a maintenance inhaler for respiratory conditions such as asthma
  Arms: Budesonide-formoterol
Drug: Placebo — Practice inhaler primarily used in training scenarios so looks identical to medical inhalers
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the impact inhalers have on blood vessels in young healthy individuals. The main question it aims to answer is if long term use of asthma inhalers have any effect on the blood vessels and heart. Participants will be asked to:

* Perform lung function and exercise tests
* Have ultrasound images taken of the artery in their arm
* Use an inhaler for 4 weeks
* Visit the lab for testing on 4-6 different occasions

Researchers will compare two different inhalers (Ventolin and Symbicort) with a placebo to see if the inhalers have any effect on the blood vessels over the 4 week period.

DETAILED DESCRIPTION:
Session 1) The first visit is a screening visit where participants will be invited to our Clinical Sciences Building research lab to conduct pulmonary function testing and cardiopulmonary exercise testing. A small blood sample will be collected via finger prick to measure hemoglobin. The cardiopulmonary screening will ensure no underlining health problems are observed in the participant which would exclude them from the study. This visit will take ~2 hours.

Session 2) The second visit will occur within 1 week of the first visit. On the second visit, participants will arrive fasted (12 hours) and be asked not to consume caffeine or perform exercise 8 hours prior to arriving. These restrictions ensure accuracy in our measurement of vascular reactivity. Measurement of cardiovascular function using heart rate, blood pressure, flow-mediated dilation, and pulse wave velocity after 10 minutes of supine rest will occur. Participants will be randomized to one of three study arms: 1) salbutamol (2x200mcg), 2) budesonide-formoterol (1x400mcg), or 3) placebo (2x0mcg). Upon receiving their group allocation, an unblinded member of the research team will help the participant in taking the required dosage, and then the participant will return to 10 minutes of supine rest. Heart rate, blood pressure, flow-mediated dilation, and pulse wave velocity will then be re-evaluated by a blinded member of the research team. Session 2 should take approximate ~1.5 hours.

Session 2A) Participants will be asked to sign a second, optional, informed consent form outlining the additional measures, techniques, and risks that are associated with the protocol. Participants will rest in the supine position and have an intravenous line inserted into the cubital fossa of the forearm. A small amount of blood will be pulled for sex hormone analysis. A 3-lead electrocardiogram will be attached, and finger blood pressure will be monitored beat-by-beat. Cardiac output will be estimated using cardiac ultrasound, while brachial blood flow will be estimated using doppler ultrasound. Muscle sympathetic nervous activity will be measured in the peroneal nerve using microneurography. Lung diffusing capacity and its components will be evaluated by standardized breath-hold techniques. In short, participants inhale a very small amount of carbon monoxide and methane and hold their breath for 6 seconds before rapidly exhaling . This maneuver is completed three times using 21%, 40%, and 60% oxygen concentration to determine diffusing capacity and pulmonary vascular function. After obtaining baseline measures of all outcomes, a beta-agonist (isoproterenol) will be injected through the intravenous line at a starting dosage of 0.01 μg∙kg-1∙min-1 for 10 minutes and increase in a stepwise manner at a rate of 0.01 μg∙kg-1∙min-1 every 10 minutes to a maximal rate of 0.04 μg∙kg-1∙min-1. The incremental dosages creating a dose-response curve for the variables blood pressure, heart rate, cardiac output, and brachial blood flow with a reduced curve indicating less β-receptor sensitivity. All values will be obtained within the last two minutes of the 10-minute dosage. Lung diffusing capacity will be evaluated following the final dosage of isoproterenol. Upon completion of infusion and data acquisition, participants will remain resting until blood pressure and heart rate return to baseline values. This session will be completed within 2 weeks of session 1 and will take ~2 hours.

Intervention: Following either session 2 or 2A if the participant consented to the additional testing session, participants will then be sent home with their inhaler and dosage regimen and complete the intervention for 4-weeks, filling out questionnaires to monitor symptoms each week. Inhalers will be equipped with electronic trackers to calculate the number of doses the participants have received.

Session 3) Following the 4-week intervention, participants will then replicate session 1 with a pulmonary function test and exercise test spanning ~2 hours. As completed during the first session, a small blood sample will be collected via finger prick to measure hemoglobin. This session will occur within 1-2 days of completing the 4-week intervention.

Session 4) Participants will be asked to arrive fasted (12 hours) and be asked not to consume caffeine or perform exercise 8 hours prior to arriving. The session will consist of the same measurements (pulse wave velocity, blood pressure, heart rate, and flow-mediated dilation) and procedure as Session 2 and spanning ~1.5 hours. This session will occur between 2-4 days following the intervention.

Session 4A) Those partaking in the additional optional visits would also then complete visit 4A which would be the same protocol as visit 2A and take ~2 hours to complete. This session will occur 3-6 days following intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18-40 years free from a medical history of cardiopulmonary disease

Exclusion Criteria:

* Absolute contraindication to exercise testing or an orthopedic condition that may limit exercise testing as identified by standardized health screening tool (PAR-Q+).
* Abnormal findings during the pulmonary function test and/or cardiopulmonary exercise test including pulmonary function values below the lower limit of normal, decrease in FEV1 following exercise (>10%), tachycardia (>100bpm at rest), and resting hypertension (>140/90 mmHg).
* Pre-existing cardiac conditions (heart failure, congenital heart defect, valvular disease) that may limit exercise testing.
* Comorbidities such as diabetes, dyslipidemia, liver disease, neuromuscular disease, renal disease, and respiratory disease
* Prescription of medical inhaler
* History of inhalants usage for greater than 1 year including but not limited to cigarettes, marijuana, and vaporizers.
* Pregnancy or lactation
* Women of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy throughout the study. Acceptable methods of contraception include tubal ligation, oral contraceptive, and barrier methods. Abstinence is an acceptable form of contraception, only insofar as patients agree to use another acceptable method of birth control, preferably a barrier method, if they become sexually active.
* Medication usage of monoamine oxidase inhibitors, tricyclic antidepressants, beta-blockers, diuretics, digoxin, other inhaled sympathomimetric bronchodilators or epinephrine, ritonavir, ketoconazole, itraconazole, cytochrome P450 sA4 inhibitors, xanthine derivatives, steroids, non-potassium sparing diuretics, L-Dopa, L-thyroxine, and oxytocin.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | Up to 3 days following intervention completion
  Velocity of blood flow between pulse points
% Increase in Brachial Artery Diameter (Flow Mediated Dilation (FMD)) | Up to 3 days following intervention completion
  Brachial artery dilation following suprasystolic occlusion

SECONDARY OUTCOMES:
Muscle sympathetic nerve activity | Up to 5 days following intervention completion
  Burst frequency of sympathetic nerve following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Bryan, MD, Study Director — University of Alberta; Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No